CLINICAL TRIAL: NCT02966106
Title: The Antidepressive Effect of Low Frequency Right Prefrontal Repetitive Transcranial Magnetic Stimulation as add-on to Antidepressant Drug Treatment. A Blinded, Placebo Controlled Randomised Study.
Brief Title: The Antidepressant Efficacy of Low Frequency rTMS as add-on
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study design was not compatible with recruiting patients to the investigation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMB-TMS-16
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2016-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right prefrontal low frequency rTMS. (Active Comparator): Right prefrontal low frequency rTMS (1Hz). A treatment session each day in four weeks apart from weekends. Each session is administered with 2 pulse trains of 180 sec with a 2 min interval
  Interventions: Device: Right prefrontal low frequency rTMS
- Sham-rTMS (Placebo Comparator): Right prefrontal rTMS sham treatment. A treatment session each day in four weeks apart from weekends. Each session is administered with 2 pulse trains of 180 sec with a 2 min interval
  Interventions: Other: Sham-rTMS

INTERVENTIONS:
Device: Right prefrontal low frequency rTMS — A treatment session each day in four weeks apart from weekends. Each session is administered with 2 pulse trains of 180 sec with a 2 min interval
  Arms: Right prefrontal low frequency rTMS.
Other: Sham-rTMS — Right prefrontal rTMS sham treatment. A treatment session each day in four weeks apart from weekends. Each session is administered with 2 pulse trains of 180 sec with a 2 min interval
  Arms: Sham-rTMS

SUMMARY:
rTMS has appeared a potential new non-invasive antidepressant method, which implies non-convulsive focal stimulation of the brain through a time varying magnetic field. ). Research on rTMS reports of minimal side effects of the method . The majority of clinically controlled studies have used high frequency stimulation of the left frontal cortex .

Fewer studies have used right prefrontal, which has less side effects, such as local discomfort and a lower risk of releasing epileptic seizures, than high frequency stimulation .Both stimulus models has been shown to have statistically significant antidepressant effect and recent research clearly indicates that low frequency rTMS of the right prefrontal cortex i associated with an antidepressant effect at the same level as the high frequency model. Therefore the investigators want to examine the antidepressant effect of a specific rTMS low frequency model in a clinical setting using a placebo controlled, randomized double blind design.

DETAILED DESCRIPTION:
rTMS has appeared a potential new non-invasive antidepressant method, which implies non-convulsive focal stimulation of the brain through a time varying magnetic field. ). RTMS is based on the principle of electromagnetism. An electromagnetic coil placed on the scalp produces a time-varying magnetic field that penetrates the scalp and skull unattenuated and gives rise to a current in the proximity of the cerebral cortex as well as functionally connected parts of the brain. Research on rTMS reports of minimal side effects of the method Previous research indicates that the antidepressant effect of rTMS is associated with specific stimulation of the dorsolateral prefrontal cortex. The stimulus frequency has shown to play a key role in the mechanisms of action of rTMS. Previous animal studies have shown that low frequency rTMS is associated with long term inhibition of neuronal activity (long term depression), while high frequency stimulation is followed by prolonged activation (long term potentiation). To some extent, this differential effect of different frequencies is reflected in human studies (REF).

The majority of clinically controlled studies have used high frequency stimulation of the left frontal cortex , which has been approved by the USA FDA (1) and later in EU for the treatment of depression.

Fewer studies have used right prefrontal, which has less side effects, such as local discomfort and a lower risk of releasing epileptic seizures, than high frequency stimulation . In addition low frequency rTMS is generally less time-consuming. Both stimulus models has been shown to have a modest, statistically significant antidepressant effect and recent research clearly indicates that low frequency rTMS of the right prefrontal cortex i associated with an antidepressant effect at the same level as the high frequency model. The issue indicates that low frequency due to the more advantagous side effect profile should be the stimulus model of choice in a clinical setting.

Therefore the investigators want to examine the antidepressant effect of a specific rTMS low frequency model in a clinical setting using a placebo controlled, randomized double blind design.

ELIGIBILITY:
Inclusion Criteria:

1. Out-patients referred to Aarhus University Hospital, Risskov
2. Moderate-severe uni- and bipolar depression according to ICD-10
3. Age 18-80 years

Exclusion Criteria:

1. Organic brain disease.
2. Epileptic seizure < 2 years
3. Patients with implanted metal parts in the brain or chest
4. Patients with pacemaker
5. Medical diseases with cerebral impact
6. Serious suicidal danger

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
remission | 8 weeks
  the number of patients obtaining a Hamilton-17 item total score of < 8

SECONDARY OUTCOMES:
Response | 8 weeks
  the number of patients obtaining a reduction in the 17-item score on the Hamilton scale for depression of >= 50%
Cognitive function | 8 weeks
  Psychological testing of cognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: Poul Erik Buchholtz, MD, Principal Investigator — Aarhus University Hospital, Risskov

IPD SHARING:
Plan to Share IPD: No